# COMPOUND AUTHORIZATION AND CONSENT FOR PARTICIPATION IN A RESEARCH PROJECT 200 FR. 1 (2016-2)

#### YALE UNIVERSITY SCHOOL OF PUBLIC HEALTH

**Study Title:** FACT-AD Study

**Principal Investigator:** Joan Monin, PhD **Funding Source:** *National Institute on Aging* 

# **Invitation to Participate and Description of Project**

We are inviting you to participate in a research study to learn about the experiences of adult children and their parents with early stage memory loss. You have been asked to participate because you have early stage memory loss. Two hundred parent-child pairs will participate in the study.

In order to decide whether or not you wish to be a part of this research study you should know enough about its risks and benefits to make an informed decision. This consent form gives you detailed information about the research study, which a member of the research team will discuss with you. This discussion should go over all aspects of this research: its purpose, the procedures that will be performed, any risks of the procedures, possible benefits and possible alternative treatments. Once you understand the study, you will be asked if you wish to participate; if so, you will be asked to sign this form.

#### **Description of Procedures**

If you agree to participate in this study, we will ask you to complete four virtual visits (by phone or computer). At the first virtual visit, you and your adult child will complete separate and private interviews that ask you questions about your health, well-being, and your relationship. After a two-week period, we will ask you to participate in a second virtual visit and participate in a series of activities and discussions in which you will be asked to talk about your experience with memory loss and other aspects of your relationship with your child on the phone or videochat. This session will be recorded. One year later, you and your child repeat theinterview visit and the activity visit again.

During the course of the study, you can continue with any other treatments you are currently receiving.

You will be told of any significant new findings that are developed during the course of your participation in this study that may affect your willingness to continue to participate. Research

l

results will not be returned to your doctor. If research results are published, your name and other personal information will not be given.

# Review of Hospital and or Office visit Records

To make sure you are suitable for this study, we will review your hospital and/or office visit records. We will use this information to check your medical history.

## **Risks and Inconveniences**

It is possible that completing interviews and talking about concerns about memory loss may cause some distress.

Other risks from participating in the study include the breach of confidentiality about your health status and participation in the study. This is very unlikely to occur, as all study investigators are trained and certified in research privacy.

## **Benefits**

Completing interviews and having discussions about concerns about your memory loss may help provide insight that may improve your well-being and relationship.

## **Economic Considerations**

The study is provided to you free of charge. There are no costs associated with your participation in the study. To thank you for participation, we will pay you in increments: \$50 for virtual visit 1, \$100 for virtual visit 2, \$50 for virtual visit 3, and \$100 for virtual visit 4.

You are responsible for paying state, federal, or other taxes for the payments you receive for being in this study. Taxes are not withheld from your payments.

#### **Treatment Alternatives/Alternatives**

If you choose not to participate in this study, there are no alternative treatments available, except those that are already being administered by your physician including pharmacotherapy (medications/drugs), exercise plans, and psychological treatments. You may choose not to participate.

## **Confidentiality and Privacy**

Any identifiable information that is obtained in connection with this study will remain confidential and will be disclosed only with your permission or as required by U.S. or State law. Examples of information that we are legally required to disclose include abuse of a child or elderly person, or certain reportable diseases. Information will be kept confidential by using only identification numbers on study forms, storing signed forms in locked cabinets, and password protecting data stored on a computer and a secure Yale data storage server. When the results of the research are published or discussed in conferences, no information will be included that

would reveal your identity unless your specific permission for this activity is obtained.

We understand that information about your health is personal, and we are committed to protecting the privacy of that information. If you decide to be in this study, the researcher will get information that identifies your personal health information. This may include information that might directly identify you, such as your name and address, telephone number, and email address, or mobile phone number. This information will be de-identified at the earliest reasonable time after we receive it, meaning we will replace your identifying information with a code that does not directly identify you. The principal investigator will keep a link that identifies you and your coded information, and this link will be kept secure and available only to the principal investigator or selected members of the research team. Any information that can identify you will remain confidential. Information will be kept confidential by using only identification numbers on study forms, storing signed forms in locked cabinets, and password protecting data stored on a computer and a secure Yale data storage server. The research team will only give this coded information to others to carry out this research study. The link to your personal information will be kept for 5 years, after which time the link will be destroyed and the data will become anonymous. The data will be kept in this anonymous form indefinitely.

### What Information Will You Collect About Me in this Study?

The information we are asking to use and share is called "Protected Health Information." It is protected by a federal law called the Privacy Rule of the Health Insurance Portability and Accountability Act (HIPAA). In general, we cannot use or share your health information for research without your permission. If you want, we can give you more information about the Privacy Rule. Also, if you have any questions about the Privacy Rule and your rights, you can speak to Yale Privacy Officer at 203-432-5919.

The specific information about you and your health that we will collect, use, and share includes:

- Research study records including recorded phone or video-chat sessions.
- Medical records held by Yale New Haven Health System or your Primary Care Provider to confirm your diagnosis for enrolling in the study, including memory loss.

Information about your health which might identify you may be used by or given to:

- The U.S. Department of Health and Human Services (DHHS) agencies
- Representatives from Yale University, the Yale Human Research Protection Program and the Yale Human Subjects Committee (the committee that reviews, approves, and monitors research on human subjects), who are responsible for ensuring research compliance. These individuals are required to keep all information confidential.
- Those individuals at Yale who are responsible for the financial oversight of research including billings and payments
- The Principal Investigator (Dr. Joan Monin)
- Co-Investigators and other investigators
- Study Coordinator and Members of the Research Team

By signing this form, you authorize the use and/or disclosure of the information described above for this research study. The purpose for the uses and disclosures you are authorizing is

to ensure that the information relating to this research is available to all parties who may need it for research purposes.

This research is covered by a Certificate of Confidentiality from the National Institutes of Health. The researchers with this Certificate may not disclose or use information, documents, or biospecimens that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other action, suit, or proceeding, or be used as evidence, for example, if there is a court subpoena, unless you have consented for this use. Information, documents, or biospecimens protected by this Certificate cannot be disclosed to anyone else who is not connected with the research except, if there is a federal, state, or local law that requires disclosure (such as to report child abuse or communicable diseases but not for federal, state, or local civil, criminal, administrative, legislative, or other proceedings, see below); if you have consented to the disclosure, including for your medical treatment; or if it is used for other scientific research, as allowed by federal regulations protecting research subjects.

The Certificate cannot be used to refuse a request for information from personnel of the United States federal or state government agency sponsoring the project that is needed for auditing or program evaluation by the National Institute on Aging which is funding this project or for information that must be disclosed in order to meet the requirements of the federal Food and Drug Administration (FDA). You should understand that a Certificate of Confidentiality does not prevent you from voluntarily releasing information about yourself or your involvement in this research. If you want your research information released to an insurer, medical care provider, or any other person not connected with the research, you must provide consent to allow the researchers to release it.

The Certificate of Confidentiality will not be used to prevent disclosure as required by federal, state, or local law of elder abuse and neglect, or harm to self or others.

The Certificate of Confidentiality will not be used to prevent disclosure for any purpose you have consented to in this informed consent document (your responses to the self-report surveys and the recoded phone or video-chat sessions).

This authorization to use and disclose your health information collected during your participation in this study will never expire.

# **Voluntary Participation and Withdrawal**

You are free to choose not to participate in this study. Your health care outside the study, the payment for your health care, and your health care benefits will not be affected if you do not agree to participate. However, you will not be able to enroll in this research study and will not receive study procedures as a study participant if you do not allow use of your information as part of this study. You do not give up any of your legal rights by signing this form.

Because this study depends on interaction between the dyad members (parent and child), if one member of the dyad wishes to withdraw, participation of the other dyad member will be terminated

# **Withdrawing From the Study**

You are free to stop and withdraw from this study at any time during its course.

To withdraw from the study, you can call a member of the research team at any time and tell them that you no longer want to take part. This will cancel any future appointments.

If you choose not to participate or if you withdraw it will not harm your relationship with your own doctors or with the Yale School of Medicine and Yale New-Haven Hospital.

## Withdrawing Your Authorization to Use and Disclose Your Health Information

You may withdraw or take away permission to use and disclose your health information at any time. You do this by calling or sending written notice to the Principal Investigator, Dr. Joan Monin Department of Social and Behavioral Sciences, Yale School of Public Health, 60 College Street, New Haven, CT 06520.

When you withdraw your permission, no new health information identifying you will be gathered after that date. Information that has already been gathered may still be used and given to others until the end of the research study, as necessary to insure the integrity of the study and/or study oversight.

# You do not give up any of your legal rights by signing this form.

#### **Ouestions**

We have used some technical terms in this form. Please feel free to ask about anything you don't understand and to consider this research and the permission form carefully – as long as you feel is necessary – before you make a decision.

## **Authorization**

I have read (or someone has read to me) this form and have decided to participate in the project described above. Its general purposes, the particulars of my involvement and possible hazards and inconveniences have been explained to my satisfaction. My signature also indicates that I have received a copy of this consent form.

| Name of Subject | et: |
|-----------------|-----|
| Signature: | |
| Date: | |

#### APPROVED BY THE YALE UNIVERSITY IRB 7/6/2022

HIC # 2000024219

| Signature of Principal Investigator | Date |
|---------------------------------------|----------|
| or | |
| Signature of Person Obtaining Consent | <br>Date |

If you have further questions about this project or if you have a research-related problem, you may contact the Principal Investigator, Dr. Joan Monin at 203 785 2895.

If, after you have signed this form you have any questions about your privacy rights, please contact the Yale Privacy Officer at 203-432-5919. If you would like to talk with someone other than the researchers to discuss problems, concerns, and questions you may have concerning this research, or to discuss your rights as a research subject, you may contact the Yale Human Subjects Committee at (203) 785-4688.